CLINICAL TRIAL: NCT06671093
Title: Phase 1b Multicenter, Open-Label Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Tune-401 in Participants With Chronic Hepatitis B Infection
Brief Title: Phase 1b, Open-label Study of Tune-401 to Assess Safety, PK and PD in Adults With Chronic Hepatitis B
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tune Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Tune-401-001
Record Dates: First submitted 2024-10-28; First posted 2024-11-04 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Chronic Hep B; Chronic Hepatitis b; Chronic Hepatitis; HBV
Keywords: Tune-401; Tune-401-001; CHB
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tune-401 Part I : Single Ascending Dose (Experimental): Epigenetic gene silencing system delivered by lipid nanoparticles (LNPs) for intravenous (IV) administration
  Interventions: Genetic: Tune-401
- Tune-401 Part II :Single/Finite Multiple Dose (Experimental): Epigenetic gene silencing system delivered by lipid nanoparticles (LNPs) for intravenous (IV) administration
  Interventions: Genetic: Tune-401

INTERVENTIONS:
Genetic: Tune-401 — Epigenetic gene silencing therapy

SUMMARY:
This study will be conducted to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of Tune-401 in adult participants with Chronic Hepatitis B.

DETAILED DESCRIPTION:
This study consists of an open-label, Part I single-ascending dose phase and Part II single and finite multiple dose phase to characterize the activity of Tune-401 on PD parameters and obtain safety data.

ELIGIBILITY:
Inclusion Criteria:

* M/F, BMI ≥ 18.5 kg/m² at screening, age 18-75, inclusive
* Diagnosed with Chronic Hepatitis B
* On nucleos(t)ide analogue
* HBeAg-negative or positive

Exclusion Criteria:

* ALT/ AST ≥ 1.5 × upper limit of normal (ULN) and total bilirubin ≥ 1. 5 × ULN
* Participants with any evidence or history of liver disease of non-HBV etiology
* Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2028-06-28 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by treatment emergent adverse events | 20 weeks
  Number of participants with treatment-related adverse events (TEAEs)

SECONDARY OUTCOMES:
Long-term safety | 104 weeks
  Number of participants with TEAEs ( safety laboratory tests (hematology, biochemistry, coagulation parameters, and urinalysis) and vital signs of clinical significance)
Tune-401 Pharmacokinetics (Cmax) | 8 weeks
  Maximum concentration (Cmax)
Tune-401 Pharmacokinetics (Tmax) | 8 weeks
  Time it takes to reach Cmax (Tmax)
Tune-401 Pharmacokinetics (AUC) | 8 weeks
  Extrapolated area under the concentration-time curve (AUC-infinity)
Tune-401 Pharmacokinetics (CL) | 8 weeks
  Clearance (CL)
Tune-401 Pharmacokinetics (half-life) | 8 weeks
  Terminal half-life (t½)
Tune-401 Pharmacokinetics (Vd) | 8 weeks
  Volume of distribution (Vd)
Tune-401 Pharmacodynamics | 104 weeks
  Changes from baseline in HBsAg
Tune-401 Immunogenicity | 104 weeks
  Development of anti-Tune-401 antibodies

CONTACTS AND LOCATIONS:
Locations (3):
- Queen Mary Hospital, University of Hong Kong, Hong Kong, Hong Kong
- PMSI Republican Clinical Hospital "Timofei Mosneaga", Arensia Exploratory Medicine Phase I Unit, Chisinau, Moldova
- New Zealand Clinical Research, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No